CLINICAL TRIAL: NCT05707546
Title: Knowledge, Beliefs and Attitudes of Greek Physiotherapists About Motivational Interviewing, Shared Decision Making and Empathetic Communication With Chronic Musculoskeletal Patients
Brief Title: Knowledge, Beliefs and Attitudes of Greek Physiotherapists About Communication With Chronic Musculoskeletal Patients
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantina Savvoulidou, Principal Investigator, University of Thessaly
Other Study IDs: N6
Record Dates: First submitted 2023-01-20; First posted 2023-02-01 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Musculoskeletal Pain; Chronic Pain
Keywords: empathy; shared decision making; motivational interviewing; physiotherapy; chronic musculoskeletal patients
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of current research study is to assess physiotherapists's knowledge, beliefs and attitudes about empathy, motivational interviewing and shared decision making in chronic musculoskeletal patients. An e-survey study will be conducted based on Checklist for Reporting Results of 52 Internet E-Surveys (CHERRIES)

DETAILED DESCRIPTION:
The main questions it aims to answer are:

What physiotherapists know about the use of empathy, motivational interviewing and shared decision making? What beliefs do physiotherapists have about the appropriate use of communication skills? Whether and how much they use empathy, motivational interview, shared decision-making in clinical practice? What are the main barriers of using communication skills (empathy, motivational interview, joint decision-making) in clinical practice?

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists who are member of Panhellenic Association of Physiotherapist in Greece, with active clinical practice in Greece and clinical experience in musculoskeletal disorders (>12 months).

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physiotherapists with chronic musculoskeletal experience and clinical practice in Greece
Sampling Method: Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Demographic characteristics | Baseline
  Questions will include participants' demographic characteristics (e.g. gender, age), 2) the setting where they practice their profession (e.g. hospital, private physiotherapy clinic), 3) level of education (e.g. BSc, MSc), 5) their years of practice, 6) seminars or training programs they have attended regarding pain neuroscience education.
Knowledge about Empathy | Baseline
  A structure questionnaire will be used which included
  1. A question about how much do they know about empathetic behaviour, using a 10-point Likert scale (0=I don't know anything about the empathetic behaviour and 10=I have comprehensive knowledge on the empathetic behaviour)"
  2. Toronto Composite Empathy Scale. The scale contains 26 statements scored on the Likert Scale (1=never, 2=sometimes, 3=less than half the time, 4=more than half the time, 5=almost all times, and 6=always). The scale demonstrated acceptable validity and reliability. The overall reliability analysis of the TCES questionnaire in Greek is high (Cronbach's α = 0.895, Sig. from Hotelling's T-Squared Test < 0.000).
Beliefs about Empathy | Baseline
  Question about how much do they believe the empathetic behaviour is useful in the treatment of chronic musculoskeletal patients, using a 6-point Likert scale (0=completely disagree and 10=completely agree).
Attitude about Empathy | Baseline
  A question about the using of the empathetic behaviour in the treatment of chronic musculoskeletal patients, using a 6-point Likert scale (0=completely disagree and 10=completely agree).
Barriers about Empathy | Baseline
  9 statements with specific barriers of showing empathy in the treatment of chronic musculoskeletal patients, using a 6-point Likert scale, where 0=completely disagree and 10=completely agree and an open question about other barriers.
Knowledge about Shared-Decision Making | Baseline
  A structure questionnaire will be used which included
  1. A question about how much do they know about the using of Shared-Decision Making, using a 10-point Likert scale (0=I don't know anything about this concept and 10=I have comprehensive knowledge about this concept)"
  2. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). The scale demonstrated acceptable validity and reliability, a Cronbach's alpha of 0.938 in the test sample.
Beliefs about Shared-Decision Making | Baseline
  A question about how much do they believe Shared-Decision Making is useful in the treatment planning of chronic musculoskeletal patients, using a 6-point Likert scale (0=completely disagree and 10=completely agree).
Attitude about Shared-Decision Making | Baseline
  A question about the using of Shared-Decision Making in the treatment planning of chronic musculoskeletal patients, using a 6-point Likert scale (0=completely disagree and 10=completely agree).
Barriers about Shared-Decision Making | Baseline
  5 statements with specific barriers of using Shared-Decision Making in the treatment planning of chronic musculoskeletal patients, using a 6-point Likert scale, where 0=completely disagree and 10=completely agree and an open question about other barriers.
Knowledge about Motivational Interviewing | Baseline
  A structure questionnaire will be used which included
  1. A question about how much do they know about the using of Motivational Interviewing, using a 10-point Likert scale (0=I don't know anything about this concept and 10=I have comprehensive knowledge about this concept)"
  2. The Motivational Interviewing Knowledge and Attitudes Test The Motivational which included true/false statements assessing knowledge of motivational interviewing principles and attitudes associated with behaviour change and the statements will be adapted for chronic musculoskeletal patients.
Beliefs about Motivational Interviewing | Baseline
  A question about how much do they believe Motivational Interviewing is useful in the treatment of chronic musculoskeletal patients, using a 6-point Likert scale (0=completely disagree and 10=completely agree).
Attitude about Motivational Interviewing | Baseline
  A question about the using of Motivational Interviewing in the treatment of chronic musculoskeletal patients, using a 6-point Likert scale (0=completely disagree and 10=completely agree).
Barriers about Motivational Interviewing | Baseline
  5 statements with specific barriers of using Motivational Interviewing in the treatment of chronic musculoskeletal patients, using a 6-point Likert scale, where 0=completely disagree and 10=completely agree and an open question about other barriers.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Kapreli, PhD, Study Director — University of Thessaly
Locations (1):
- University of Thessaly, Lamia, Greece

IPD SHARING:
Plan to Share IPD: Undecided